CLINICAL TRIAL: NCT06833541
Title: Research on Gut-kidney Axis Regulation of Diabetic Kidney Disease Based on Multi-omics and Bacterio-drug Interaction Control Mechanism
Brief Title: Research on Gut Microbiota and Metabolomics in Diabetic Kidney Disease
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: U21A20411
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Nephropathy Type 2; Type 2 Diabetes Mellitus (T2DM); Chronic Kidney Disease
Keywords: Diabetic Nephropathy Type 2; Type 2 diabetes mellitus; chronic kidney disease; intestinal microbiota; metabolomics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, urine supernatant, feces, tongue coating
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Type 2 Diabetes Kidney Disease: Clinical diagnostic criteria consistent with Type 2 Diabetes Kidney Disease
- Type 2 Diabetes Mellitus: Clinical diagnostic criteria consistent with Type 2 Diabetes Mellitus(T2DM)
- Chronic Kidney Disease: Clinical diagnostic criteria consistent with Chronic Kidney Disease (CKD)
- healthy people: Relatively healthy people without diabetes and chronic kidney disease

SUMMARY:
Diabetic kidney disease (DKD) is characterized by high prevalence, multiple pathogenesis, and lack of effective treatment and management strategies. Early detection helps overcome treatment inertia, enables timely medical intervention, maximizes renal function in diabetic patients, and is essential to avoid renal failure and improve clinical outcomes. The gold standard for diagnosis of DKD is renal biopsy, which has the highest accuracy. However, due to the trauma of renal biopsy, the patient acceptance is low, the application scenario is not universal, and it is only used when it is difficult to distinguish diabetic nephropathy from non-diabetic nephropathy, and it is not the preferred diagnostic method for DKD.

In the past decade, with the emergence and application of metabonomics, proteomics, genomics and other multi-omics techniques, more and more studies have recognized the prominent role of intestinal flora disorders and gut-derived metabolites in the occurrence of DKD. Therefore, from the perspective of intestinal flora, using multi-omics techniques to identify enterogenic metabolic markers of DKD and restore intestinal flora balance may be potential strategies for prevention and management of DKD. Modern medicine believes that intestinal flora is not only closely related to diet and digestion, participating in the synthesis, absorption and metabolism of nutrients, but also constituting intestinal barrier and participating in immune defense of the body. Its function is similar to the physiological function of "The spleen governs transportation and transformation".

Based on the traditional Chinese medicine（TCM） pathogenesis of DKD "Spleen Failure to Disperse Essence and Poison Damage Kidney Collateral" proposed by the previous research group, this study intends to use microbiology-metabolomics to deeply study the TCM pathogenesis of DKD, provide scientific basis for it, and guide the theory of traditional Chinese medicine widely used in clinical work of prevention and treatment of diabetic nephropathy.

DETAILED DESCRIPTION:
This study is a single-center, parallel trial design. It is prepared to recruit subjects with type 2 diabetes kidney disease (DKD), Type 2 diabetes mellitus(T2DM), chronic kidney disease (CKD), and healthy individuals based on clinical diagnostic criteria and screening criteria. While observing main indicators such as blood glucose, glycosylated hemoglobin, and renal function, blood, urine, feces, and tongue coating samples are collected and frozen. The 16S rDNA technology, metagenomics technology, targeted and non-targeted metabolomics technology are used to detect the results and analyze the differences. Subsequently, based on the detection results, 4-6 remaining fecal samples from each group will be selected as human-intestinal flora donors for "human-germ-free mouse" faecal microbiota transplantation.

ELIGIBILITY:
Patient inclusion criteria：

1. Age ≥18 years old and ≤75 years old, gender is not limited.
2. Complete demographic data.
3. Meet the diagnostic criteria of the Chinese Guidelines for the Prevention and Treatment of Diabetic Kidney Disease (2021 edition), the Chinese Guidelines for the Prevention and Treatment of Type 2 Diabetes Mellitus (2020 edition), and the Guidelines for the Screening, Diagnosis, Prevention and Treatment of Chronic Kidney Disease (2017 edition).
4. The patient is informed of the study as approved by the ethics committee.

Healthy population inclusion criteria:

(1) The patient has no known history of infection or risk factors including HIV hepatitis B or C virus syphilis etc. and no current systemic infection; (2) No obesity (body mass index >30) and/or diabetes no history of chronic kidney disease; (3) Approved by the ethics committee patients were informed about the study. Exclusion criteria：

1. A history of infection or other acute disease within one month prior to enrollment.
2. Current state of stress.
3. Other unstable chronic diseases;
4. A history of acute and chronic gastrointestinal diseases, including acute gastroenteritis, functional gastrointestinal diseases, inflammatory bowel disease, celiac disease, and other chronic gastrointestinal diseases.
5. Individuals who have received systemic antibiotics, immunosuppressants, chemotherapy, or chronic treatment with proton pump inhibitors within the past three months will be excluded from participation.
6. Pregnant or lactating women will also be excluded.
7. Individuals who have participated in other drug clinical trials within the past three months will be excluded.
8. Individuals who suffer from mental illness, intellectual disability, confusion, or other conditions that may interfere with their ability to cooperate with the completion of relevant information collection will also be excluded.

Those who were unable to cooperate with the collection of pertinent data were likewise excluded from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients are treated at the Department of Endocrinology or the Department of Nephrology in the First Affiliated Hospital of Hunan University of Traditional Chinese Medicine, and those who meet the inclusion criteria. At the same time, healthy people who meet the inclusion criteria are recruited through recruitment advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 720 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
UACR | Complete once at enrollment
  Urine Albumin-to-Creatinine Ratio
eGFR | Complete once at enrollment
  Estimated Glomerular Filtration Rate
BUN | Complete once at enrollment
  blood urea nitrogen
Scr | Complete once at enrollment
  serum creatinine
FBG | Complete once at enrollment
  fasting blood glucose
HbA1c | Complete once at enrollment
  Glycosylated Hemoglobin, Type A1C
GSP | Complete once at enrollment
  glucosylated serum protein

SECONDARY OUTCOMES:
16S rDNA | Complete once at enrollment
  16S ribosomal DNA identification
Targeted Metabolomics | Complete once at enrollment
  Targeted Metabolomics technology detection
Non-targeted metabolomics | Complete once at enrollment
  Non-targeted metabolomics technology detection
mNGS | Complete once at enrollment
  metagenomic Next Generation Sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Juan Huang, Doctor, Principal Investigator — The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine; Rong Yu, Doctor, Study Director — The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine
Locations (1):
- The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT06833541/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT06833541/ICF_001.pdf